CLINICAL TRIAL: NCT05953402
Title: ZEPOSIA® (Ozanimod) Ulcerative Colitis Pregnancy Registry: a Prospective, Observational Study on the Safety of Ozanimod Exposure in Pregnant Women With Ulcerative Colitis and Their Offspring
Brief Title: A Study of Ozanimod in Pregnant Women With Ulcerative Colitis and Their Offspring
Status: Not yet recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-026
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
Keywords: ZEPOSIA®; Ozanimod; Pregnancy; Sphingosine-1-phosphate (S1P) therapies; Inflammatory Bowel Disease; IBD; Ulcerative Colitis; UC
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months

GROUPS / COHORTS (3):
- Ozanimod-exposed participants with UC: Pregnant women with a diagnosis of UC who are exposed to ozanimod at any time during pregnancy
- Conventional therapy-exposed participants with UC: Pregnant women with a diagnosis of UC who are exposed to conventional therapies (aminosalicylates and/or thiopurines) but not exposed to ozanimod, other S1P therapies, or advanced therapies for UC (biologics and/or small molecules) at any time during pregnancy
- Advanced therapy-exposed participants with UC: Pregnant women with a diagnosis of UC who are exposed to advanced therapies for UC (biologics and/or small molecules) but not exposed to ozanimod or other S1P therapies at any time during pregnancy

SUMMARY:
The purpose of this study is to evaluate association between ozanimod exposure during pregnancy and subsequent maternal, fetal, and infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently or recently pregnant
* Diagnosis of UC
* Resident of country where ozanimod is prescribed for the treatment of UC

Exclusion Criteria:

* Exposure to other S1P therapies at any time during pregnancy

Other protocol-defined eligibility criteria apply.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include women of any age who i) are currently or recently have been pregnant; ii) have a diagnosis of UC; iii) reside in a country where ozanimod is prescribed for the treatment of UC; iv) provide consent to participate as well as medical releases for their Healthcare Providers (HCPs) to provide data to the registry; and v) meet the criteria for inclusion.
Sampling Method: Probability Sample
Enrollment: 1182 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2033-06-29 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Event rate of Major Congenital Malformations (MCM) | Up to 12 months

SECONDARY OUTCOMES:
Event rate of minor congenital malformations | Up to 12 months
Event rate of pre-eclampsia | Up to 9 months
Event rate of eclampsia | Up to 9 months
Event rate of Spontaneous Abortion (SAB) | Up to 9 months
Event rate of stillbirth | Up to 9 months
Event rate of elective termination | Up to 9 months
Event rate of preterm birth | Up to 9 months
Event rate of Small for Gestational Age (SGA) | Up to 12 months
Event rate of postnatal growth deficiency | Up to 12 months
Event rate of infant developmental deficiency | Up to 12 months
Event rate of perinatal death | Up to 10 months
Event rate of neonatal death | Up to 1 month
Event rate of infant death | Up to 12 months
Event rate of serious or opportunistic infant infections | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm